CLINICAL TRIAL: NCT03323437
Title: Biomarkers of Conversion Risk and Treatment Response in Early-Stage Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York State Psychiatric Institute (Other); Columbia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1702018001; R01MH110270 (NIH)
Record Dates: First submitted 2017-10-02; First posted 2017-10-27 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patient (Experimental): Medication-free individuals during first-episode of psychosis who will receive 4 weeks of treatment with risperidone
  Interventions: Drug: Risperidone
- Control (No Intervention): Healthy, psychosis-free controls who will not receive risperidone

INTERVENTIONS:
Drug: Risperidone — Participants will meet with a study doctor physician once per week (about 3 times total) to monitor progress and side-effects of risperidone, which includes taking 4 assessments each time. After 4 weeks of taking Risperidone, participant will be assessed and scanned with the MRI/MRS scanner again.
  Arms: Patient

SUMMARY:
Schizophrenia (SZ) is a highly debilitating neuropsychiatric disorder of young adulthood onset and a leading cause of disability worldwide. While treatments delivered at early stages of the disorder may be effective at reducing psychosis or altering the course of the disease, there are currently no biomarkers capable of identifying subjects in early stages of SZ who are likely to respond to treatment and would be good candidates for available proactive, symptomatic or future disease-modifying treatments; or those who would not respond and can be spared unnecessary medication exposure. The lack of these vitally important biomarkers provides a compelling rationale for the present multidisciplinary research project, which aims to develop and validate highly promising noninvasive and objective proton magnetic resonance spectroscopy (1H MRS)-based biomarkers for monitoring treatment response in early stages of SZ. In support of the viability of this overall objective is a large body of data, reported by the applicants and others, that show (a) that levels of glutamate (Glu) and - aminobutyric acid (GABA) - respectively, the major excitatory and inhibitory amino acid neurotransmitter systems - are abnormally elevated in medication-naïve and unmedicated first episode and chronic SZ patients; (b) that the effect of treatment with antipsychotic medications in these populations may be to lower or normalize brain levels of both Glu and GABA. To investigate the potential of these in vivo brain Glu and GABA abnormalities to serve as biomarkers of treatment response in early-stage SZ, the applicants propose to use 1H MRS to measure Glu and GABA levels in the largest cohort of medication-free SZ subjects to date, at baseline and following 4 weeks of antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria (Patients):

1. Male or females between the ages of 18-35
2. less than five years (<60 months) of active Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
3. Capacity to provide informed consent
4. No major medical or neurological illness
5. Medication free (3 weeks without antipsychotic medications)

Exclusion Criteria (Patients):

1. Current alcohol or drug abuse (<1 month) or substance dependence (<6 months) or substances used within one day of the imaging study.
2. Pregnant or lactating women or women of child-bearing potential, who are either not surgically-sterile or, for outpatients, not using appropriate methods of birth control.
3. Intelligence Quotient (IQ) <70
4. Acute risk for suicide or violence
5. Presence of pacemaker or any metallic objects in the body that would interfere with the MRS or cause MRI safety problems
6. Claustrophobia
7. Any organic brain disorder (including epilepsy, mental retardation, or a medical condition whose pathology or treatment would likely alter the presentation or treatment of SZ
8. Individuals on anti-epileptic medications (e.g., valproate, carbamazepine) that may affect GABA or Glu
9. Unstable medical or neurological condition
10. DSM-V diagnosis of bipolar disorder I
11. DSM-V diagnosis of major depression with psychotic features
12. History of non-response to or non-tolerance of Risperidone

Inclusion Criteria (Healthy Controls)

1. Male or females between the ages of 18-35
2. less than five years (<60 months) of active DSM diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
3. No major medical or neurological illness

Exclusion Criteria (Healthy Controls)

1. Current alcohol or drug abuse (<1 month) or substance dependence (<6 months) or substances used within one day of the imaging study.
2. Pregnant or lactating women or women of child-bearing potential, who are either not surgically-sterile or, for outpatients, not using appropriate methods of birth control.
3. IQ<70
4. Acute risk for suicide or violence
5. Presence of pacemaker or any metallic objects in the body that would interfere with the MRS or cause MRI safety problems
6. Claustrophobia
7. History of psychotropic medication use such as antipsychotics or antidepressants
8. Any first-degree family history of psychotic illness
9. Personal history of any DSM Axis I disorder
10. Individuals on anti-epileptic medications (e.g., valproate, carbamazepine) that may affect GABA or Glu
11. Unstable medical or neurological condition
12. Any organic brain disorder (including epilepsy, mental retardation, or a medical condition whose pathology or treatment would likely alter the presentation or treatment of SZ

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dikoma C. Shungu, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York State Psychiatric Institute & Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abi-Dargham A, Gil R, Krystal J, Baldwin RM, Seibyl JP, Bowers M, van Dyck CH, Charney DS, Innis RB, Laruelle M. Increased striatal dopamine transmission in schizophrenia: confirmation in a second cohort. Am J Psychiatry. 1998 Jun;155(6):761-7. doi: 10.1176/ajp.155.6.761. PMID 9619147
- [Background] Carlsson A, Waters N, Holm-Waters S, Tedroff J, Nilsson M, Carlsson ML. Interactions between monoamines, glutamate, and GABA in schizophrenia: new evidence. Annu Rev Pharmacol Toxicol. 2001;41:237-60. doi: 10.1146/annurev.pharmtox.41.1.237. PMID 11264457
- [Background] CARLSSON A, LINDQVIST M. EFFECT OF CHLORPROMAZINE OR HALOPERIDOL ON FORMATION OF 3METHOXYTYRAMINE AND NORMETANEPHRINE IN MOUSE BRAIN. Acta Pharmacol Toxicol (Copenh). 1963;20:140-4. doi: 10.1111/j.1600-0773.1963.tb01730.x. No abstract available. PMID 14060771
- [Background] Coyle JT. The glutamatergic dysfunction hypothesis for schizophrenia. Harv Rev Psychiatry. 1996 Jan-Feb;3(5):241-53. doi: 10.3109/10673229609017192. PMID 9384954
- [Background] Davis KL, Kahn RS, Ko G, Davidson M. Dopamine in schizophrenia: a review and reconceptualization. Am J Psychiatry. 1991 Nov;148(11):1474-86. doi: 10.1176/ajp.148.11.1474. PMID 1681750
- [Background] Farooq S, Large M, Nielssen O, Waheed W. The relationship between the duration of untreated psychosis and outcome in low-and-middle income countries: a systematic review and meta analysis. Schizophr Res. 2009 Apr;109(1-3):15-23. doi: 10.1016/j.schres.2009.01.008. Epub 2009 Feb 23. PMID 19233621
- [Background] Fusar-Poli P, Bonoldi I, Yung AR, Borgwardt S, Kempton MJ, Valmaggia L, Barale F, Caverzasi E, McGuire P. Predicting psychosis: meta-analysis of transition outcomes in individuals at high clinical risk. Arch Gen Psychiatry. 2012 Mar;69(3):220-9. doi: 10.1001/archgenpsychiatry.2011.1472. PMID 22393215
- [Background] Fusar-Poli P, Borgwardt S, Bechdolf A, Addington J, Riecher-Rossler A, Schultze-Lutter F, Keshavan M, Wood S, Ruhrmann S, Seidman LJ, Valmaggia L, Cannon T, Velthorst E, De Haan L, Cornblatt B, Bonoldi I, Birchwood M, McGlashan T, Carpenter W, McGorry P, Klosterkotter J, McGuire P, Yung A. The psychosis high-risk state: a comprehensive state-of-the-art review. JAMA Psychiatry. 2013 Jan;70(1):107-20. doi: 10.1001/jamapsychiatry.2013.269. PMID 23165428
- [Background] Javitt DC, Zukin SR. Recent advances in the phencyclidine model of schizophrenia. Am J Psychiatry. 1991 Oct;148(10):1301-8. doi: 10.1176/ajp.148.10.1301. PMID 1654746
- [Background] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Background] Lodge DJ, Grace AA. Aberrant hippocampal activity underlies the dopamine dysregulation in an animal model of schizophrenia. J Neurosci. 2007 Oct 17;27(42):11424-30. doi: 10.1523/JNEUROSCI.2847-07.2007. PMID 17942737
- [Background] Laruelle M, Abi-Dargham A. Dopamine as the wind of the psychotic fire: new evidence from brain imaging studies. J Psychopharmacol. 1999 Dec;13(4):358-71. doi: 10.1177/026988119901300405. PMID 10667612
- [Background] Laruelle M, Abi-Dargham A, van Dyck CH, Gil R, D'Souza CD, Erdos J, McCance E, Rosenblatt W, Fingado C, Zoghbi SS, Baldwin RM, Seibyl JP, Krystal JH, Charney DS, Innis RB. Single photon emission computerized tomography imaging of amphetamine-induced dopamine release in drug-free schizophrenic subjects. Proc Natl Acad Sci U S A. 1996 Aug 20;93(17):9235-40. doi: 10.1073/pnas.93.17.9235. PMID 8799184
- [Background] Moghaddam B, Adams B, Verma A, Daly D. Activation of glutamatergic neurotransmission by ketamine: a novel step in the pathway from NMDA receptor blockade to dopaminergic and cognitive disruptions associated with the prefrontal cortex. J Neurosci. 1997 Apr 15;17(8):2921-7. doi: 10.1523/JNEUROSCI.17-08-02921.1997. PMID 9092613
- [Background] Olney JW, Farber NB. Glutamate receptor dysfunction and schizophrenia. Arch Gen Psychiatry. 1995 Dec;52(12):998-1007. doi: 10.1001/archpsyc.1995.03950240016004. PMID 7492260
- [Background] Olsen KA, Rosenbaum B. Prospective investigations of the prodromal state of schizophrenia: review of studies. Acta Psychiatr Scand. 2006 Apr;113(4):247-72. doi: 10.1111/j.1600-0447.2005.00697.x. PMID 16638070
- [Background] Perkins DO, Gu H, Boteva K, Lieberman JA. Relationship between duration of untreated psychosis and outcome in first-episode schizophrenia: a critical review and meta-analysis. Am J Psychiatry. 2005 Oct;162(10):1785-804. doi: 10.1176/appi.ajp.162.10.1785. PMID 16199825
- [Background] Snyder SH. The dopamine hypothesis of schizophrenia: focus on the dopamine receptor. Am J Psychiatry. 1976 Feb;133(2):197-202. doi: 10.1176/ajp.133.2.197. PMID 1251927
- [Background] Tamminga CA. Schizophrenia and glutamatergic transmission. Crit Rev Neurobiol. 1998;12(1-2):21-36. doi: 10.1615/critrevneurobiol.v12.i1-2.20. PMID 9444480
- [Background] Tamminga CA, Holcomb HH, Gao XM, Lahti AC. Glutamate pharmacology and the treatment of schizophrenia: current status and future directions. Int Clin Psychopharmacol. 1995 Sep;10 Suppl 3:29-37. PMID 8866763
- [Background] Yung AR, Yuen HP, Berger G, Francey S, Hung TC, Nelson B, Phillips L, McGorry P. Declining transition rate in ultra high risk (prodromal) services: dilution or reduction of risk? Schizophr Bull. 2007 May;33(3):673-81. doi: 10.1093/schbul/sbm015. Epub 2007 Apr 2. PMID 17404389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient | Control
Started | 13 | 13
Completed | 13 | 9
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: There are only 9 control subjects in the overall number of baseline participants as 4 of the 13 control subjects who were eligible decided to withdraw before completing the baseline procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient | Control | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (3.3) | 26.4 (2.7) | 24.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Biomarkers of Treatment Response: Dorsal Caudate (DCA) Gamma Amino Butyric Acid (GABA) Levels
Description: Dorsal Caudate (DCA) GABA levels will be ascertained at baseline and after 4 weeks of treatment using MRI scan with 1H MRS to assess treatment response. This is a measure of GABA levels, over water, in the dorsal caudate. For patients this is a change measure. For control subjects, this is a one time measure. The values can range from 0 to infinity for controls and -infinity to infinity for patients.
Time Frame: Baseline and 4 weeks of treatment for patients, baseline for controls
Population: The number of participants analyzed is lower than the participant flow as data from several subjects were excluded due to MRS quality control issues brought about by unreliable performance of a head coil.
Measure: Mean (95% Confidence Interval); unit: institutional units
Arm/Group | Patient | Control
Number analyzed (Participants) | 10 | 8
institutional units | -0.65 [-0.95 to -0.35] | .0037 [.00333 to .0040]
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p < 0.01, ANOVA

2. Primary Outcome: Change in Biomarkers of Treatment Response: Dorsal Caudate (DCA) Glx (Glutamate+Glutamine)
Description: Dorsal Caudate (DCA) Glx levels will be ascertained at baseline and after 4 weeks of treatment using MRI scan with 1H MRS to assess treatment response. This is a measure of the levels of Glx over water in the dorsal caudate. For patients this is a change measure. For control subjects, this is a one time measure. The values can range from 0 to infinity for controls and -infinity to infinity for patients.
Time Frame: Baseline and 4th week of treatment for patients, baseline only for controls
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: institutional units
Arm/Group | Patient | Control
Number analyzed (Participants) | 10 | 8
institutional units | -.28 [-.80 to 0.24] | .00221 [.00198 to .00244]
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .68, ANOVA

3. Primary Outcome: Change in Biomarkers Reflecting Treatment Response: Medial Prefrontal Cortex (MPFC) Gamma Amino Butyric Acid (GABA)
Description: Medial Prefrontal Cortex (MPFC) GABA levels will be ascertained at baseline and after 4 weeks of treatment using MRI scan with 1H MRS to assess treatment response. This is a measure of GABA levels, over water, in the mPFC. For patients this is a change measure. For control subjects, this is a one time measure. The values can range from 0 to infinity for controls and -infinity to infinity for patients.
Time Frame: Baseline and 4th week of treatment for patients, baseline only for controls
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: institutional units
Arm/Group | Patient | Control
Number analyzed (Participants) | 10 | 8
institutional units | .85 [.05 to 1.64] | .00247 [.0022 to .0025]
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .03, ANOVA

4. Primary Outcome: Change in Biomarkers Reflecting Treatment Response: Medial Prefrontal Cortex (MPFC) Glx (Glutamate+Glutamine)
Description: Medial Prefrontal Cortex (MPFC) Glx levels will be ascertained at baseline and after 4 weeks of treatment using MRI scan with 1H MRS to assess treatment response. This is a measure of glx levels, over water, in the mPFC. For patients this is a change measure. For control subjects, this is a one time measure. The values can range from 0 to infinity for controls and -infinity to infinity for patients.
Time Frame: Baseline and 4th week of treatment for patients, baseline for controls
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: institutional units
Arm/Group | Patient | Control
Number analyzed (Participants) | 10 | 8
institutional units | 0.19 [-.54 to .93] | .00191 [.00174 to .00208]
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .01, ANOVA

5. Secondary Outcome: Changes in Neurocognitive Performance: MATRICS Consensus Cognitive Battery (MCCB)
Description: Memory, attention, reasoning, emotional intelligence, and verbal ability will be assessed using the MCCB before and after 4 weeks of treatment. MATRICS Consensus Cognitive Battery (MCCB) as measure of Neurocognitive/Functional Measures is a standardized battery designed to measure cognitive functioning in people with schizophrenia. The MCCB is represented as a percentile score. This score can go from 0 to 100 where a higher score indicates a better performance. For patients this is a change measure. For control subjects, this is a one time measure.
Time Frame: Baseline and 4th week of of treatment for patients, baseline only for controls
Population: The number of participants analyzed is lower than the participant flow as some subjects did not finish all assessments in the MATRICS necessary to calculate this outcome.
Measure: Mean (Full Range); unit: percentile score
Arm/Group | Patient | Control
Number analyzed (Participants) | 8 | 8
percentile score | 0.222 [0 to 34.4] | 42.9 [1.4 to 91.9]
Statistical Analysis 1: Comparison: Patient; Test type: Other — two sided t test; p = .59, t-test, 2 sided

6. Secondary Outcome: WAMI (Wealth Asset and Income)
Description: The WAMI Score at Baseline is a measure of socioeconomic status across countries and culture. The index scale goes from 0 (lower socioeconomic situation) to 1 (highest socioeconomic situation).
Time Frame: Baseline
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Control
Number analyzed (Participants) | 7 | 5
score on a scale | .901 (.179) | .982 (.027)
Statistical Analysis 1: Comparison: Patient vs Control; Test type: Other — two sided t test; p = .45, t-test, 2 sided

7. Secondary Outcome: Changes in Clinical Symptomatology: Positive and Negative Syndrome Scale (PANSS)
Description: Changes in Positive and Negative Symptoms will be assessed across the treatment period using the PANSS.
  Participants are rated on a scale of
  1. (Absent)
  2. (Minimal)
  3. (Mild)
  4. (Moderate)
  5. (Moderate severe)
  6. (Severe)
  7. (Extreme)
  to describe Positive, Negative and General symptomatology. Items from each subscale (Positive, Negative, and General) are summed for their respective scales, with lower numbers indicating less severe or absent symptomatology, and higher scores indicating more severe symptoms. A total sum of all subscales is also computed to reflect overall symptom severity.
  Positive Subscale: 7 items, minimum score = 7, maximum score = 49 Negative Subscale: 7 items, minimum score = 7, maximum score = 49 General Subscale: '16 items, minimum score = 16, maximum score = 112 Total Score: 30 items, minimum score = 30, maximum score = 210.
  For patients this is a change measure. For control subjects, this is a one time measure.
Time Frame: Baseline and week 4 for patients; for controls only baseline
Population: The number of participants analyzed is lower than the participant flow as some subjects were unable to complete all measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Control
Number analyzed (Participants) | 12 | 9
score on a scale | -0.09 (.15) | 31.89 (2.98)
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .32, ANOVA

8. Secondary Outcome: Changes in Motor Symptomatology: Abnormal Involuntary Movement Scale (AIMS)
Description: Motor symptomatology associated with tardive dyskinesia (TD) assessed using the AIMS.
  The measure consists of 10 items with scale/scores for each item of:
  0 None
  1. Minimal
  2. Mild
  3. Moderate
  4. Severe Higher ratings = higher levels of motor symptoms which is worse. This scale assesses abnormal movements for parts of the body.
  The total score is a sum score of items 1-10 and can be 0-40, with 40 being the most symptomatic (i.e., most extrapyramidal side effects, or worse).
Time Frame: Baseline and week 4
Population: This measure is solely for patients and people who received antipsychotic treatment, so control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient
Number analyzed (Participants) | 13
score on a scale | -.077 (.28)
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .60, ANOVA

9. Secondary Outcome: Changes in Clinical Severity: Clinical Global Impression Scale
Description: Changes in clinical severity over the course of treatment will be monitored using the The Clinical Global Impression Scale (CGI) consists of two items.- Severity scale (CGI-S).
  Severity - The first item assesses the patient's current level of mental health symptomatology compared to the clinician's experience with other patients with the same diagnosis. The scale ranges from
  1. (Normal, not at all ill)
  2. (Borderline mentally ill)
  3. (Mildly ill)
  4. (Moderately ill)
  5. (Markedly ill)
  6. (Severely ill)
  7. (Among the most extremely ill patients)
  Improvement - The second item assesses how much the patient's symptomatology has changed since the last clinical visit.
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
  For patients this is a change measure. For control subjects, this is a one time measure.
  The possible score range is 1-7 with 1 being least and 7 being most symptomatic.
Time Frame: Baseline and week 4 for patients; for controls this is a baseline measure only
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete all measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Control
Number analyzed (Participants) | 13 | 9
score on a scale | -0.054 (.10) | 1 (0)
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .34, ANOVA

10. Secondary Outcome: Changes in Global Functioning: Global Assessment of Functioning (GAF)
Description: Changes in global functioning over the course of treatment will be assessed using the Global Assessment of Functioning (GAF).
  Participants are rated 1-100 on their level of functioning, according to clinical observation:
  91 - 100 No symptoms. 81 - 90 Absent or minimal symptoms 71 - 80 If symptoms are present, they expected reactions to stressors 61 - 70 Some mild symptoms 51 - 60 Moderate symptoms 41 - 50 Serious symptoms 31 - 40 Impairment in reality testing or communication or major impairment in several areas 21-30 Behavior influenced by delusions or hallucinations or serious impairment in communication/judgment/inability to function in almost all areas 11-20 Some danger of hurting self or others or occasionally fails to maintain minimal personal hygiene or gross impairment in communication 1-10 Persistent violence risk or lack of self-care 0 No info
  For patients this is a change measure. For control subjects, this is a one time measure.
Time Frame: Baseline and week 4 for patients; for controls only baseline
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Control
Number analyzed (Participants) | 12 | 9
score on a scale | 0.21 (.20) | 86.4 (8.53)
Statistical Analysis 1: Comparison: Patient; Test type: Other — two way anova; p = .35, ANOVA

11. Secondary Outcome: Recreational Substances Used by Patients as Recorded by the Substance Use Questionnaire
Description: This measure is a self-reported questionnaire which assesses for any use of the following substances within the past month prior to the initial research visit Tobacco (if the respondent indicates that they have used tobacco in the past month, they are additionally asked, "On average, how many cigarettes per day have you smoked in the past 7 days?" Alcohol, Cocaine, Marijuana, Opiates, Amphetamines, phencyclidine (PCP) Other Drugs of Abuse (if the respondent indicates they have used other drugs of abuse within the past month of the initial research visit, they are given the opportunity to "specify" which other drugs of abuse they used
Time Frame: This measure is administered on Day 1 of the study.
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete all measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient | Control
Number analyzed (Participants) | 10 | 9
Participants | 6 | 4
Statistical Analysis 1: Comparison: Patient vs Control; Test type: Other — fisher's exact; p = .66, Fisher Exact

12. Secondary Outcome: Participants' Verbal I.Q (Intelligence Quotient) as Assessed by the WTAR (Wechsler Test of Adult Reading) to Determine Clinical Eligibility
Description: This measure assesses a participant's verbal ability to determine whether they are cognitively able to complete the measures involved in the study. The participant will read from a list of 50 English words and the rater will record whether the pronunciation was correct on a score card for each word spoken. A standard score below the 70th percentile on this measure is indicative of an intellectual disability which would exclude a participant from being clinically and cognitively eligible to complete this study. The potential score range is 0-50. A higher score indicates better cognitive ability. There is only one total score.
Time Frame: This measure is completed on Day 1 of the study.
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete all measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient | Control
Number analyzed (Participants) | 14 | 9
score on a scale | 36.9 (8.43) | 43.9 (6.23)
Statistical Analysis 1: Comparison: Patient vs Control; Test type: Other — two sided t test; p = .04, t-test, 2 sided

13. Secondary Outcome: Participants' Self-Reported Handedness as Recorded by the Edinburgh Handedness Scale (Predominantly Right)
Description: This measure assesses a participant's preference regarding which hand they would use to complete a specific task. They have the option to indicate whether they would use they would always or most of the time use their left, right, or both left and right hands to complete each task. This measure assesses handedness based on the amount of responses which indicate the participant is either left handed, right handed, or ambidextrous. Below we specifically report on the number of individuals who were predominantly right handed.
Time Frame: This measure is completed on Day 1 of the study.
Population: The number of participants analyzed is lower than the participant flow as some subjects did not complete all measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient | Control
Number analyzed (Participants) | 13 | 9
Participants | 11 | 7
Statistical Analysis 1: Comparison: Patient vs Control; Test type: Other — fisher's exact test; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: 4-6 weeks for patients, 1-2 weeks for controls
Arm/Group | Patient | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 12/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient (N=13) | Control (N=13)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
restlessness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
drowsiness/sedation (Nervous system disorders) | 8 (10) | 0 (0)
involuntary movements (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03323437/Prot_SAP_000.pdf